CLINICAL TRIAL: NCT02709070
Title: Resection Combined With Highly-purified CTL Versus Resection Alone for HCC
Brief Title: Resection+Highly Purified CTL Versus Resection Alone for HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, MD.PhD., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 005
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: highly-purified CTL
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- resection (Active Comparator): Resection was carried out under general anesthesia using a right subcostal incision with a midline extension. Intra-operative ultrasonography was performed routinely to evaluate the tumor burden, liver remnant and the possibility of a negative resection margin. The investigators performed anatomical resection aiming at a resection margin of at least 1 cm. Pringle's maneuver was routinely used with a clamp and unclamp time of 10 minutes and 5 minutes, respectively. Hemostasis of the raw liver surface was done with suturing and application of fibrin glue.
  Interventions: Procedure: resection
- highly-purified CTL (Experimental): Peripheral blood (20-30mL) for manufacturing the individualized highly-purified CTL agent was collected from the respective participants who were randomized to the immunotherapy group before starting treatment. The highly-purified CTL agent was prepared at a central manufacturing facility. Participants in the immunotherapy group received a number up to 5×10E9 of the highly-purified CTL agent intravenously over 60 minutes without any premedication and then were observed for at least 30 minutes. Participants were scheduled to receive highly-purified CTL: 4-6 treatments at a frequency of once two-week during 6 months after receiving resection, followed by 6-9 treatments during 6 months to 2 years after receiving resection.
  Interventions: Procedure: resection; Procedure: highly-purified CTL

INTERVENTIONS:
Procedure: resection — hepatectomy for HCC
Procedure: highly-purified CTL — hepatectomy first, followed by highly-purified CTL treatment
  Arms: highly-purified CTL

SUMMARY:
There is little evidence showed that adjuvant therapy had been shown to extend the survival of patients with hepatocellular carcinoma (HCC) receiving surgical resection. We investigated whether injections of highly-purified Cytotoxic T lymphocytes prolongs recurrence-free survival of patients after resection for HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common and the third leading cause of cancer-related death worldwide. Resection is considered as the main curative treatment for HCC, but recurrence of tumor within the liver remnant is common, with a reported 5-year recurrence rate of 70%, which results in poor prognosis of HCC, and the high recurrence rate has led efforts to develop adjuvant therapies to reduce recurrence. However, the benefit of any form of adjuvant therapy remains unclear. Current guidelines didn't recommend any adjuvant therapy after resection. A previous clinical trial from Japan reported that cytokine-induced killer(CIK) cell immunotherapy increased recurrence-free survival (RFS) after surgical resection of HCC. Immunotherapy has become an optional treatment for HCC. Cytotoxic T lymphocytes(CTL), a kind of effective T cells that specific recognizing and killing antigen targeted cells through cloning amplification after receiving antigen information from antigen presented cell and playing key role to clear cancerous cells. There is little evidence for adjuvant CTL treatment for HCC receiving resection. So our hypothesis is that adjuvant highly-purified CTL is superior to resection alone for HCC. The aim of this prospective study is to compare the outcome of resection combined with highly-purified CTL with resection for HCC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years; 2. First diagnosed HCC, no other treatment received; 3.Child-pugh A-B 4. No severe coagulation disorders (prothrombin activity<40% or a platelet count<40,000/mm3); 5. Eastern Co-operative Oncology Group performance(ECOG) status 0-1.

Exclusion Criteria:

* 1. Pregnant women, breastfeeding women or plan pregnancy for the future 2 years; 2. The presence of vascular invasion or extrahepatic spread on imaging; 3. Usage of strong immunosuppressive agents such as corticosteroids, cyclosporine A within six months or longer; 4. HIV antibody or hepatitis C virus antibody positive; 5. Immunodeficiency diseases or autoimmune diseases (such as rheumatoid arthritis, Buerger's disease, multiple sclerosis and type 1 diabetes); 6. Suffering with cancers (except skin cancer, prostate cancer or cervical carcinoma in situ) at the enrolling time or 5 years before; 7. Suffering with other organ failure; 8. Suffering with severe mental illness; 9. Drug addiction (including alcohol) for 1 year before the enrolling time; 10. Participate in other Clinical trials within three months prior to 3 months before the enrolling time; 11. Other researchers believe that the patient is not fit for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
recurrence free survival | 2-year
  from the date of randomization to the first recurrence or to death from any cause

SECONDARY OUTCOMES:
overall survival | 5-year
  from the date of randomization until death from any cause, and cancer-specific survival was measured from the date.
  from the date of randomization until death from any cause, and cancer-specific survival was measured from the date of randomization until death resulting from HCC

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lee JH, Lee JH, Lim YS, Yeon JE, Song TJ, Yu SJ, Gwak GY, Kim KM, Kim YJ, Lee JW, Yoon JH. Adjuvant immunotherapy with autologous cytokine-induced killer cells for hepatocellular carcinoma. Gastroenterology. 2015 Jun;148(7):1383-91.e6. doi: 10.1053/j.gastro.2015.02.055. Epub 2015 Mar 4. PMID 25747273
- [Background] Peng ZW, Zhang YJ, Chen MS, Xu L, Liang HH, Lin XJ, Guo RP, Zhang YQ, Lau WY. Radiofrequency ablation with or without transcatheter arterial chemoembolization in the treatment of hepatocellular carcinoma: a prospective randomized trial. J Clin Oncol. 2013 Feb 1;31(4):426-32. doi: 10.1200/JCO.2012.42.9936. Epub 2012 Dec 26. PMID 23269991
- [Background] Takayama T, Sekine T, Makuuchi M, Yamasaki S, Kosuge T, Yamamoto J, Shimada K, Sakamoto M, Hirohashi S, Ohashi Y, Kakizoe T. Adoptive immunotherapy to lower postsurgical recurrence rates of hepatocellular carcinoma: a randomised trial. Lancet. 2000 Sep 2;356(9232):802-7. doi: 10.1016/S0140-6736(00)02654-4. PMID 11022927